CLINICAL TRIAL: NCT03413254
Title: Second and Third Look Laparoscopy in pT4 Colon Cancer Patients for Early Detection of Peritoneal Metastases; the COLOPEC-II Randomized Multicentre Trial
Brief Title: Second and Third Look Laparoscopy in pT4 Colon Cancer Patients for Early Detection of Peritoneal Metastases
Acronym: COLOPEC-II
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, P.J. Tanis, M.D. PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL61507.018.17
Record Dates: First submitted 2018-01-05; First posted 2018-01-29 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer; Peritoneal Metastases
Keywords: pT4 colon cancer; Peritoneal metastases; Early detection; Diagnostic laparoscopy; Second look surgery; Third look surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Masking Description: In order to prevent caretakers from being influenced by the assigned follow-up strategy, the randomization outcome will remain unknown to everyone involved in the patient's care until the 18 months CT-scan is reported by the radiologist.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2nd look DLS + routine FU (Active Comparator): Follow-up after curatively resected pT4 colon cancer, consisting of second look DLS after negative CT abdomen at 6-9 months and normal CEA, with subsequent routine follow-up according to the Dutch colorectal cancer guideline until 5 years.
  Interventions: Other: Routine follow-up; Procedure: Second look DLS
- 2nd and 3rd DLS + routine FU (Experimental): Follow-up after curatively resected pT4 colon cancer, consisting of second look DLS after negative CT abdomen at 6-9 months and normal CEA, with subsequent routine follow-up and third look DLS after negative CT abdomen at 18 months and normal CEA. Third look DLS is not performed in patients with evidence of disease that is not curable, or in those already diagnosed with PM in the preceding period.
  Interventions: Other: Routine follow-up; Procedure: Second look DLS; Procedure: Third look DLS

INTERVENTIONS:
Other: Routine follow-up — Patients visit the outpatient clinic twice a year during the first two to three years and annually thereafter, until five years postoperative. CEA-levels are determined at 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 48 and 60 months after primary resection. Detection of liver metastases with ultrasound or CT is performed at 12, 24, 36, 48 and 60 months postoperative. At 6 and 18 months postoperative, a CT-scan is part of the study protocol, but ultrasound of the liver is allowed for other time intervals during follow-up. Colonoscopy is performed at 12 and 48 months postoperative.
Procedure: Second look DLS — Second look DLS is performed within one month from negative CT at 6-9 months (depending last date of adjuvant chemotherapy) and normal CEA. Laparoscopic access to the abdominal cavity is obtained under general anaesthesia, followed by adhesiolysis if necessary. Complete staging is performed, with biopsy of any lesion suspicious of PM, and determining the peritoneal cancer index (PCI) in case of PM. Conversion to laparotomy not allowed for better exposure, but only for intra-operative complications.
Procedure: Third look DLS — Third look DLS is performed within one month from negative CT at 18 months and normal CEA. Laparoscopic access to the abdominal cavity is obtained under general anaesthesia, followed by adhesiolysis if necessary. Complete staging is performed, with biopsy of any lesion suspicious of PM, and determining the peritoneal cancer index (PCI) in case of PM. Conversion to laparotomy not allowed for better exposure, but only for intra-operative complications.
  Arms: 2nd and 3rd DLS + routine FU

SUMMARY:
The COLOPEC II multicentre randomized trial will investigate the role of second and third look laparoscopy to detect metachronous peritoneal metastases at a clinically occult stage during the follow-up of pT4 colon cancer patients. It is expected that detection of PM at a clinically occult stage will translate into survival benefit, due to higher percentage of patients eligible for curative intent treatment with cytoreductive surgery (CRS) and hyperthermic intraperitoneal chemotherapy (HIPEC).

DETAILED DESCRIPTION:
Problem description Approximately 20-30% of patients with pT4 colon cancer develop peritoneal metastases (PM). The only proven curative option for macroscopic PM is cytoreductive surgery (CRS) followed by hyperthermic intraperitoneal chemotherapy (HIPEC), but the efficacy and morbidity highly depend on the extent of peritoneal involvement. Unfortunately, due to restricted accuracy of imaging modalities and the absence of early symptoms, PM are often detected at a stage in which only about 20-25% of patients are eligible for CRS+HIPEC, and even these patients appear to have a relatively high peritoneal cancer index (PCI). New diagnostic strategies are urgently required to detect PM at an early stage, resulting in a higher percentage of patients eligible for CRS+HIPEC, which will translate into better survival because of the uniformly reported direct association between PCI and survival.

Proposed solution Preliminary findings of the COLOPEC trial (NCT02231086) revealed that PM were already detected at intentionally adjuvant HIPEC within 2 months after resection of the primary tumour in 10% of patients with pT4 colon cancer. Based on these findings and literature, second look diagnostic laparoscopy (DLS) to detect PM when the disease is still potentially curable by CRS+HIPEC may be considered as an essential component of early follow-up of pT4 colon cancer. This needs confirmation in a larger patient cohort before implementing this in practice. Furthermore, metachronous PM develop later on (>12 months) in an additional 15-20% of the patients. These patients will be missed by a second look DLS and might therefore benefit from a third look DLS later on, which will be investigated in the COLOPEC II trial.

Objective The primary aim of this study is to determine the added value of third look DLS after a negative second look DLS in pT4 colon cancer patients to detect PM at a clinically occult stage.

Study design This is a randomized multicentre trial in which eligible patients will have routine CT-abdomen at 6 months postoperative (+3 months for those still treated with adjuvant chemotherapy), followed by second look DLS within 1 month after CT if no PM or other metastases not amenable for local treatment are detected. Patients without PM found during second look DLS will subsequently be randomized between routine follow-up including CT-abdomen at 18 months in the control arm, or an experimental arm with a third look DLS provided that PM or incurable metastases are absent at the 18 months CT-abdomen. The primary endpoint of the study is the proportion of PM detected after negative second look DLS. The primary endpoint will be determined at 20 months.

Study population Patients aged 18-80 years who underwent intentionally curative resection of pT4a,bN0-2M0 colon cancer or rectosigmoid cancer above the peritoneal reflection, either with or without adjuvant systemic chemotherapy, who are fit enough and surgically accessible to undergo second look DLS between 6-10 months postoperatively and subsequent treatment of PM if detected.

Intervention DLS will be performed in patients not already diagnosed with PM and without other metastases that impede curative intent treatment. Access to the abdominal cavity is obtained under general anaesthesia by open introduction away from areas of expected adhesions, followed by adhesiolysis if necessary. Complete staging of the intra-abdominal cavity is performed, with biopsy of any lesion suspicious of PM, and determining the PCI for those patients with suspected PM.

Expected outcome It is hypothesized that in patients who had a negative second look DLS, PM become clinically apparent in 5% until 20 months postoperatively with routine follow-up. A third look DLS following a negative CT-abdomen at 18 months postoperative is expected to detect an additional 10% of PM. It is expected that detection of PM at a clinically occult stage will translate into survival benefit, based on the observation that survival rates after CRS+HIPEC are higher if the PCI is lower.

ELIGIBILITY:
Inclusion Criteria:

* Curative intent resection of pT4a,bN0-2M0 colon cancer or rectosigmoid cancer above the peritoneal reflection, with or without adjuvant systemic therapy;
* Age between 18 and 80 years;
* Written informed consent.

Exclusion Criteria:

* Histological subtype other than (mucinous) adenocarcinoma or signet-ring cell carcinoma;
* Clinical condition that does not allow for second look surgery or subsequent treatment of PM if detected;
* Second look surgery thought not to be technically possible (i.e. because of extensive abdominal surgery / re-interventions).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of peritoneal metastases detected after a negative second look DLS | 20 months
  Peritoneal metastases that are detected using either routine follow-up or third look DLS according to randomization.

SECONDARY OUTCOMES:
Incidence of PM at second look DLS after curative treatment of primary tumour, depending on pathological pT4 stage, pathological nodal stage and histology | 6-10 months
  Occult peritoneal metastases not detected by routine CT scan 6-9 months after primary resection of pT4 colon cancer, that are detected at second look DLS performed at 6-10 months after the primary resection.
Incidence of PM during first 20 months after curative resection of primary tumour, depending on pathological pT4 stage, pathological nodal stage and histology | 20 months
  This outcome measure tries to stratify pT4 colon cancer patients in clinically relevant subgroups based on their risk to develop PM.
Incidence of PM in patients who did or did not undergo adjuvant chemotherapy | 20 months
  This outcome measure analysis a potential impact of adjuvant chemotherapy on the development of PM.
Sensitivity, specificy, NPV and PPV of CT imaging to detect PM compared to DLS | 20 months
  Diagnostic accuracy of CT using DLS findings as gold standard.
Proportion of detected PM eligible for curative intent CRS+HIPEC at different follow-up intervals | 20 months
  This outcome measures determines the clinical impact of PM detection, considering potentially curative intent treatment.
30-day morbidity related to second/third look DLS | From the second or third look DLS till 30 days postoperative
  This outcome measure is important to determine the harm/benefit ratio of DLS.
Extent of adhesiolysis required at second/third look DLS assessed with the Zühlke score | 20 months
  The Zühlke score measures the severity of intraabdominal adhesions.
  1. Filmy adhesions.
  2. Stronger adhesions requiring some sharp dissection.
  3. Dense vascularized adhesions requiring sharp dissection.
  4. Extreme dense vascularized adhesions with high risk for organ damage during dissection.
  A higher score indicates a worse outcome.
5-year peritoneal recurrence free survival | 5 years
  This outcome measure determines whether third look DLS has any impact on the overall detection of PM.
5-year disease-free survival | 5 years
  Important long-term oncological endpoint to determine the potential oncological benefit of third look DLS.
5-year overall survival | 5 years
  Important long-term oncological endpoint to determine the potential oncological benefit of third look DLS.
Quality of life assessed with the CRC-29 questionnaire | 2 years
  Assessing impact of invasive diagnostic procedures on QOL.
Quality of life assessed with the EQ-5D-5L questionnaire | 2 years
  Assessing impact of invasive diagnostic procedures on QOL.

CONTACTS AND LOCATIONS:
Locations (10):
- Netherlands (10):
  - Flevoziekenhuis, Almere Stad
  - Amsterdam UMC, location AMC, Amsterdam
  - Amsterdam UMC, location VUmc, Amsterdam
  - Antoni van Leeuwenhoek, Amsterdam
  - OLVG, Amsterdam
  - Catharina hospital, Eindhoven
  - University Medical Center Groningen, Groningen
  - St. Antonius hospital, Nieuwegein
  - Radboudumc, Nijmegen
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No